CLINICAL TRIAL: NCT04169945
Title: Subgingival Debridement by Erythritol Powder Air-Polishing (EPAP) in Comparison With Ultrasonic Instrumentation During Periodontal Maintenance. A Randomised Clinical Trial
Brief Title: Compare Air Polishing With Ultrasonic During Maintenance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Nor Adinar Baharuddin, Associate Professor, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 101269-3
Record Dates: First submitted 2019-11-14; First posted 2019-11-20 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Periodontitis
Keywords: periodontitis; air polishing; randomised clinical trial; debridement
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasonic instrumentation and Air Polishing (Experimental): All participants will receive full mouth conventional ultrasonic subgingival debridement, followed by air-polishing with erythritol powder which include activating device for 5 seconds of each surface (Petersilka 2003). Subsequently, Perio-Flow handpiece with a special disposable nozzle will be used for pocket depth >4mm. Perio-Flow handpiece with a special disposable nozzle will be used for pocket depth >4mm
  Interventions: Other: Ultrasonic instrumentation; Other: Air polishing with erythritol powder
- Ultrasonic instrumentation (Active Comparator): All participants will receive full mouth conventional ultrasonic subgingival debridement only. No time limit (Flemmig 2012), until dental surfaces feel smooth.
  Interventions: Other: Ultrasonic instrumentation

INTERVENTIONS:
Other: Ultrasonic instrumentation — Full mouth root surface debridement
Other: Air polishing with erythritol powder — Air flow PLUS
  Arms: Ultrasonic instrumentation and Air Polishing

SUMMARY:
Periodontal disease is a chronic multifactorial inflammatory disease that affects the soft and hard supporting tissues of the teeth. It is one of the most common oral health problems which 90% of the global adult population has been reported to have some form of the disease. Microorganisms in dental biofilm play a critical etiological factor in the development of this progressive destruction disease, and if left untreated, will eventually lead to tooth loss. Recurrent periodontal disease did occur in treated and well-maintained patients at different time intervals and is a site-specific disorder. Therefore, subgingival biofilm removal during supportive periodontal therapy has become a fundamental part in achieving a stable oral health after completion of active treatment. Subgingival debridement involves various techniques. In recent years, many studies have reported on the effectiveness of air polishing device using different powders versus conventional hand instruments and/or oscillating scalers. However, there is no study evaluating the health economic aspect of these treatment modalities. As development leads to advancement of treatment options, they often involve higher cost than the existing measures. Therefore, besides clinical efficacy, economic evaluation enables health decision makers to allocate limited health resources in a more efficient manner, to ensure best possible outcomes, without neglecting any segment of care.

DETAILED DESCRIPTION:
As a result of ongoing microbiological challenge from accumulated dental plaque, it is paramount to ensure thorough removal of such deposits from the root surface to maintain periodontal health. Mechanical instrumentation using conventional hand instrument and/or oscillating scalers is the gold standard of periodontal therapy. Patient is commonly recalled every 3-4 months interval for supportive periodontal therapy (SPT) to decrease disease recurrence and prevent further tooth loss. This repeated mechanical instrumentation, however, may cause irreversible damage to dental hard tissue. As such, the use of treatment modalities effective in removing biofilm, being time efficient, causing minimal discomfort, tissue damage, and less abrasion of root surface would be preferable during SPT.

With the advancement of technology in dentistry, air polishing (AP) was introduced to dentistry for cavity reparation in 1945. The usage then extended into periodontal debridement in SPT, by means of slurry pressurized air with a novel low abrasive powder and water. A study done by Petersilka et al. 2003 in 27 SPT patients of pockets 3-5mm depth revealed an approximately 90% reduction in all viable bacterial counts and offered greater patient comfort when compared to conventional hand instrument. It was also time saving as only 5 seconds is needed per tooth surface. Since 1980s, sodium bicarbonate has been used in AP devices and was the only powder available until 2004. It is non-toxic, water-soluble, safe for intra-oral use and is efficient in removing biofilm and staining on intact enamel surfaces. However, this conventional powder can cause substantial damage to the root cementum and dentine at area of receded gingiva, severe epithelial erosion and unpleasant perception by patients.

In order to deal with this issue, several types of AP abrasive powders with improved clinical performance and patient comfort have been produced. As early as in 2003, glycine based (amino acid) powders were produced with smaller mean particle size 45-60 µm and less chiseled shape, compared to sharp edged and up to 250 µm mean particle size of sodium bicarbonate. Due to its ≈80% less abrasiveness, studies had shown that glycine powder air-polishing (GPAP) was more efficient in plaque removal in root debridement, caused non-critical substance loss and lower the rate of increase in root surface roughness when compared to sodium bicarbonate. On the other hand, in a publication by Flemmig et al. in 2007, efficacy of GPAP was assessed in periodontal pockets of various depths. The results revealed the average debridement depth of 2mm was obtained at pockets depth of 4mm, and 60% of subgingival root surface was cleaned. In deeper pockets, the efficacy reduced to about 40% and the use of hand instruments or ultrasonic scalers may be superior.

Thus, Moёne et al. had described a newly designed nozzle in 2010 in order to extend the use of air polishing in deeper pockets. This nozzle allowed access to subgingival root surfaces and the jet spray has a lower flow and pressure compared to supragingivally applied air polishing. This new device appeared to be safe, perceived to be more acceptable by patients and was more time efficient than scaling and root planing. However, Petersilka (2010) pointed out two cases of air emphysema developed after using this jet system but fortunately the cases resolved within 4 days without additional intervention. Therefore, he remarked that emphysema cannot be completely ruled out in all other types of air-polishing systems. Since then, more studies have been carried out using this newly designed nozzle with GPAP. A 2-months trial by Wennstrӧm et al. in 20 recall patients showed no significant differences in clinical or microbiological outcomes between subgingivally applied GPAP (SubGPAP) and ultrasonic debridement of moderate deep pockets (5-8mm). They also noted there was only a short-term reduction of subgingival microflora in both modalities.

Recently, a natural sugar erythritol powder has gained its popularity as it has slightly lower abrasiveness and smaller particle size 14-31 µm compared to glycine. In 2013, Hashino et al. found that erythritol has inhibitory effect on the biofilm produced by Streptococcus gordonii and Porphyromonas gingivalis. A year after, Drago and team tested on a new formulation consisting of erythritol and chlorhexidine with the standard glycine powder. This in vitro study demonstrated that the combination of erythritol/chlorhexidine displayed a stronger antimicrobial and antibiofilm activity on titanium discs. While in a 12 months clinical trial by Müller and co-workers, repeated subgingival air polishing with erythritol containing 0.3% chlorhexidine appeared to be safe, reduced the number of pockets >4mm and induced less pain than ultrasonic instrumentation. As subgingival biofilm may not mineralise between two SPT visits, less aggressive approach with better microbiological outcome may be appropriate for residual pockets.

Based on the available literature, requirements like time efficiency, minimal hard and soft tissue damage, along with high patient acceptance and safety, are important for repeated treatments especially in SPT. Whether a new air-polishing powder, used with a specially designed nozzle may be a valid alternative to conventional debridement, cost efficiency is another essential aspect to be defined. As periodontitis patients need long-term professional care and in the light of rising healthcare costs, a cost- and clinically effective treatment modality is required.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 30 to 65 years old.
* Patients with at least 20 teeth available.
* Patients already in SPT at least 3 months after completion of comprehensive periodontal therapy.
* Presence of at least 4 teeth with residual pockets of ≥5mm and positive bleeding on probing.
* Patients with controlled systemic diseases.

Exclusion Criteria:

* Patients with a plaque control record >30%.
* Patients who had undergone radiation or immunosuppressive therapy.
* Patients with cardiac pacemaker, defibrillators and any implantable electronic device.
* Patients who are on antibiotics, anti-inflammatory drugs or other medication taken within the previous 3 months.
* Patients who are confirmed or suspected intolerance to the test products.
* Patients with history or known case of root hypersensitivity.
* Patients with physical limitation that might hinder proper home care or oral hygiene procedures.
* Patients who are pregnant.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Presence of pocket depth >4mm | 6 months
  To determine presence of pocket depth > 4 mm after 6 months

SECONDARY OUTCOMES:
Clinical attachment level gain (CAL) | 6 months
  To determine presence of CAL after 6 months
Patient reported outcome measures (PROM) | 6 months
  Patient reported outcome measures using visual analogue scales score where 0 is no pain and 10 is the worst pain
Incremental Cost Effectiveness Ratio (ICER) | 6 months
  Incremental Cost Effectiveness Ratio
Patient reported outcome measures (PROM) | 6 months
  Patient reported outcome measures using oral health impact profile (OHIP-14) score, based on the likert scale responses; which were coded as (1) very often, (2) quite often, (3) sometimes, (4) seldom, (5) never and (6) don't know.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drago L, Del Fabbro M, Bortolin M, Vassena C, De Vecchi E, Taschieri S. Biofilm removal and antimicrobial activity of two different air-polishing powders: an in vitro study. J Periodontol. 2014 Nov;85(11):e363-9. doi: 10.1902/jop.2014.140134. Epub 2014 Jul 25. PMID 25060742
- [Background] Flemmig TF, Petersilka GJ, Mehl A, Hickel R, Klaiber B. The effect of working parameters on root substance removal using a piezoelectric ultrasonic scaler in vitro. J Clin Periodontol. 1998 Feb;25(2):158-63. doi: 10.1111/j.1600-051x.1998.tb02422.x. PMID 9495615
- [Background] Hashino E, Kuboniwa M, Alghamdi SA, Yamaguchi M, Yamamoto R, Cho H, Amano A. Erythritol alters microstructure and metabolomic profiles of biofilm composed of Streptococcus gordonii and Porphyromonas gingivalis. Mol Oral Microbiol. 2013 Dec;28(6):435-51. doi: 10.1111/omi.12037. Epub 2013 Jul 29. PMID 23890177
- [Background] Mohd-Dom TN, Wan-Puteh SE, Muhd-Nur A, Ayob R, Abdul-Manaf MR, Abdul-Muttalib K, Aljunid SM. Cost-Effectiveness of Periodontitis Management in Public Sector Specialist Periodontal Clinics: A Societal Perspective Research in Malaysia. Value Health Reg Issues. 2014 May;3:117-123. doi: 10.1016/j.vhri.2014.04.012. Epub 2014 May 20. PMID 29702916
- [Background] Petersilka GJ, Bell M, Mehl A, Hickel R, Flemmig TF. Root defects following air polishing. J Clin Periodontol. 2003 Feb;30(2):165-70. doi: 10.1034/j.1600-051x.2003.300204.x. PMID 12622860
- [Background] Sahrmann P, Ronay V, Schmidlin PR, Attin T, Paque F. Three-dimensional defect evaluation of air polishing on extracted human roots. J Periodontol. 2014 Aug;85(8):1107-14. doi: 10.1902/jop.2014.130629. Epub 2014 Jan 30. PMID 24476548
- [Background] Wennstrom JL, Dahlen G, Ramberg P. Subgingival debridement of periodontal pockets by air polishing in comparison with ultrasonic instrumentation during maintenance therapy. J Clin Periodontol. 2011 Sep;38(9):820-7. doi: 10.1111/j.1600-051X.2011.01751.x. Epub 2011 Jul 7. PMID 21736599
- [Background] Zappa U, Smith B, Simona C, Graf H, Case D, Kim W. Root substance removal by scaling and root planing. J Periodontol. 1991 Dec;62(12):750-4. doi: 10.1902/jop.1991.62.12.750. PMID 1765938
- [Result] Buhler J, Schmidli F, Weiger R, Walter C. Analysis of the effects of air polishing powders containing sodium bicarbonate and glycine on human teeth. Clin Oral Investig. 2015 May;19(4):877-85. doi: 10.1007/s00784-014-1317-z. Epub 2014 Sep 21. PMID 25240922
- [Result] Farooqi OA, Wehler CJ, Gibson G, Jurasic MM, Jones JA. Appropriate Recall Interval for Periodontal Maintenance: A Systematic Review. J Evid Based Dent Pract. 2015 Dec;15(4):171-81. doi: 10.1016/j.jebdp.2015.10.001. Epub 2015 Nov 19. PMID 26698003
- [Result] Flemmig TF, Hetzel M, Topoll H, Gerss J, Haeberlein I, Petersilka G. Subgingival debridement efficacy of glycine powder air polishing. J Periodontol. 2007 Jun;78(6):1002-10. doi: 10.1902/jop.2007.060420. PMID 17539712
- [Result] Lindhe J, Nyman S. Long-term maintenance of patients treated for advanced periodontal disease. J Clin Periodontol. 1984 Sep;11(8):504-14. doi: 10.1111/j.1600-051x.1984.tb00902.x. PMID 6384275
- [Result] Lindhe J, Westfelt E, Nyman S, Socransky SS, Haffajee AD. Long-term effect of surgical/non-surgical treatment of periodontal disease. J Clin Periodontol. 1984 Aug;11(7):448-58. doi: 10.1111/j.1600-051x.1984.tb01344.x. PMID 6378986
- [Result] Moene R, Decaillet F, Andersen E, Mombelli A. Subgingival plaque removal using a new air-polishing device. J Periodontol. 2010 Jan;81(1):79-88. doi: 10.1902/jop.2009.090394. PMID 20059420
- [Result] Muller N, Moene R, Cancela JA, Mombelli A. Subgingival air-polishing with erythritol during periodontal maintenance: randomized clinical trial of twelve months. J Clin Periodontol. 2014 Sep;41(9):883-9. doi: 10.1111/jcpe.12289. Epub 2014 Aug 7. PMID 25041441
- [Result] Petersilka GJ, Steinmann D, Haberlein I, Heinecke A, Flemmig TF. Subgingival plaque removal in buccal and lingual sites using a novel low abrasive air-polishing powder. J Clin Periodontol. 2003 Apr;30(4):328-33. doi: 10.1034/j.1600-051x.2003.00290.x. PMID 12694431
- [Result] Petersilka GJ. Subgingival air-polishing in the treatment of periodontal biofilm infections. Periodontol 2000. 2011 Feb;55(1):124-42. doi: 10.1111/j.1600-0757.2010.00342.x. No abstract available. PMID 21134232